CLINICAL TRIAL: NCT06647771
Title: Relationship Between First 12-h Body Temperature and Acute Kidney Injury After Valvular Heart Surgery
Brief Title: Relationship Between Postoperative Tempeartive and Acute Kidney Injury
Status: Active, not recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-0771
Record Dates: First submitted 2024-10-13; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Patients Undergoing Valvular Heart Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to identify body temperature trajectory classes based on core temperature changes during the first 12 hours post-surgery and to explore their relationship with postoperative acute kidney injury in patients undergoing valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent valvular heart surgery between January 2016 and July 2023 at Severance Cardiovascular Hospital of Yonsei University Health System

Exclusion Criteria:

* Patients who underwent the same surgery within 30 days,
* Patients with less than two temperature measurements within 12 hours after surgery, - Patients with missing creatinine test values before and within seven days after surgery,
* Patients who died during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 3274 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury ≥ stage 2 according to the KDIGO criteria | seven days after valvular heart surgery
  According to the KDIGO criteria, postoperative acute kidney injury of stage 2 or higher was defined as a 100% increase in creatinine within the first seven days after surgery. The association between stage 2-3 acute kidney injury and postoperative body temperature trajectory classes was investigated.

SECONDARY OUTCOMES:
non-recovery from acute kidney injury within 48 | 72 hours after the onset of acute kidney injury
  The association between postoperative body temperature trajectory classes and non-recovery from acute kidney injury was investigated at two time points: within 48 hours
non-recovery from acute kidney injury within 72 hours | 72 hours after the onset of acute kidney injury
  The association between postoperative body temperature trajectory classes and non-recovery from acute kidney injury was investigated at two time points: within 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No